CLINICAL TRIAL: NCT03154918
Title: A Study of Gemcitabine, L- Asparaginase, Ifosfamide, Dexamethasone and Etoposide Chemotherapy Followed by ASCT for Newly Diagnosed Stage IV, Relapsed or Refractory Extranodal Natural Killer/T-cell Lymphoma, Nasal Type
Brief Title: GLIDE Regimen Followed by ASCT for Aggressive NK/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Attending Physician, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXNKT 1.0
Record Dates: First submitted 2017-05-02; First posted 2017-05-16 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — Dexamethasone; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLIDE (Experimental): Treated with GLIDE regiment chemotherapy for 4 cycles.
  Interventions: Drug: GLIDE

INTERVENTIONS:
Drug: GLIDE — The dose and schedule of GLIDE chemotherapy was as follows: gemcitabine 800 mg/m 2 days 1, 8; Peg-ASP 2500 U/m 2 days 4; ifosfamide 1000 mg/m 2 days 1 - 3; dexamethasone 20 mg days 1 - 4; etoposide 100 mg/m 2 days 1 - 3.
  Other Names: gemcitabine,Peg-ASP,ifosfamide,dexamethasone and etoposide

SUMMARY:
This study is to explore the efficacy and safety of GLIDE regiment in patients with aggressive NK/T cell lymphoma.

DETAILED DESCRIPTION:
Treatment

The dose and schedule of GLIDE chemotherapy was administered as following: gemcitabine 800 mg/m2, day 1,5; peg-asparaginase 2000 u/m2, day 4,11; ifosfamide 1000 mg/m2, day 1-3; etoposide 100mg/m2, day 1-3; dexamethasone 20mg day 1-4 . Gemcitabine on day 5 should be skipped if any grade 3 or above hematologic toxicities developed. Peg-asparaginase should be discontinued if patients developed any asparaginase related allergic reaction. Granulocyte colony stimulating factor was started on day 4 till full recovery of absolute neutrophils count (ANC, defined as above 2×109/L). The interval between 2 cycles of chemotherapy is 4 weeks and before initiation of a new cycle of chemotherapy, severity of all non-hematologic adverse events must be less than grade 2, ANC above 2×109/L and platelets count above 80×109/L. If adverse events failed to recover, the following cycle of chemotherapy should be postponed for one week. If there was no recovery 4 weeks before the day of the scheduled following cycle, the protocol treatment was terminated. Totally, 6 cycles of GLIDE chemotherapy was planned for protocol treatment. Response of lymphoma should be evaluated every 2 cycles.

Hematopoietic stem cells of patients with best response better than partial response (PR), including PR and complete response (CR) after up to 6 cycles of GLIDE, were collected. receive When complete response is attained, peripheral hematopoietic stem cells should be collected. Fitted patients will treated with chidamide, cladribine, gemcitabine and busulfan ( ChiCGB) conditioning followed by autologous stem cell transplantation (ASCT). Patients who are unable to receive ASCT, continued with GLIDE for up to 6 cycles. Patients who are unable to attain PR after 6 cycles of GLIDE, drop off this trial.

Response and Toxicity Evaluation Baseline evaluations were finished 10 days before enrollment, including history, physical examination, complete blood count, serum liver and kidney function, serum lactate dehydrogenase level, marrow smear and biopsy, enhanced computer tomography of neck, thorax, abdomen and pelvis and endoscopic investigation of gastrointestinal tract if such sites involvement were indicated. Response was regularly evaluated after every two cycles of GLIDE chemotherapy using the revised response criteria for malignant lymphoma. Therefore, in this trial, complete response (CR) was defined as the complete disappearance of all objective signs of disease, including enlarged lymph nodes or hepatomegaly and splenomegaly at the restaging. Partial response (PR) was defined as at least a 50% reduction of tumor volume without the occurrence of new lesions at the restaging. Progressive disease was defined as a greater than 25% increase in the sum of tumor lesions or the emergence of one or more new lesion(s) or clinical symptoms that indicate disease progression. No response was defined as any response that did not fall into the other defined categories. The toxicity of treatment was graded using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0.

Statistical Analysis Outcome analysis was performed using life table methods and associated statistics. The primary endpoints were ORR and CR rate after 4 cycles of GLIDE chemotherapy. The second end points were 3-year OS and toxicity. Survival estimates were calculated using the Kaplan-Meier method. All analysis were performed using Prism, version 5.0, software (Graphpad Software, Inc.)

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of ENKL defined by World Health Organization classification 2008;
2. age above 18 years;
3. Eastern Cooperative Oncology Group performance status of 0-3;
4. adequate organ function defined as: total bilirubin≤2 times the upper limit of normal; alanine aminotransferase and aspartate aminotransferase levels≤2.5 times the upper limit of normal; serum creatinine≤1.5 mg/dL; creatinine clearance ≥50 mL/minute and normal electrocardiogram results.

Exclusion Criteria:

1. uncontrolled infection;
2. pregnant or lactating women;
3. contraindication to one of the trial drugs (eg. anaphylaxis to L-asparaginase);
4. any coexisting medical problems of sufficient severity to prevent full compliance with the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 2 years after recruitment
  2-year progression free survival

SECONDARY OUTCOMES:
CR | 2 and 6 month after GLIDE, and 3 month after ASCT
  complete remission
AEs | 2 years after recruitment
  adverse events
OS | 2 years after recruitment
  2-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Ting Liu, MD, Study Director — West China Hospital
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
on-line shared files